CLINICAL TRIAL: NCT04832308
Title: Mobile Intervention Supervised Exercise Therapy Study 1
Acronym: MiSET-1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of grant funding
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Society for Vascular Surgery (Other)
Responsible Party: Principal Investigator, Oliver Aalami, Clinical Associate Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61023
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Artery Disease; Claudication, Intermittent
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Block randomization stratified by site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVS SET Program (Experimental): Participants enroll in SVS Program which includes 1) educational information on PAD, exercise and nutrition, 2) weekly health coaching, and 3) walking therapy prescription.
  Interventions: Behavioral: Exercise Therapy
- Usual Care (No Intervention): This usual care arm will allow sites to direct patients as they usually do. This could include an in-person exercise therapy program or simply exercise instruction during an office visit.

INTERVENTIONS:
Behavioral: Exercise Therapy — This is a health coach driven exercise prescription for patients recommending 30 minutes or more of moderate effort walking 3-5 days a week with expected walk-rest-walk-rest intervals.
  Arms: SVS SET Program

SUMMARY:
This is a randomized controlled trial evaluating the impact of the mobile phone delivered SVS SET Program on utilization, functional capacity, symptoms and quality of life.

DETAILED DESCRIPTION:
This is a national randomized controlled study with approximately 10-15 sites enrolling patients with Rutherford II peripheral artery disease (PAD) in total. Patients will be randomized between the SVS SET Program and "usual care" for each site. The primary outcome will be to study the site-specific effect on utilization of exercise therapy. Secondary outcomes will be the effect on the 6-minute-walk test, passive activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of Age
* Rutherford Class I-II PAD (claudication)
* Ambulatory
* Exercise Therapy Naive (>18 mo)
* Primary Owner of an Android or iOS device
* Willingness to participate (text, call, fill out surveys) via a mobile phone

Exclusion Criteria:

* Symptomatic coronary artery disease
* Oxygen dependent COPD
* Significant osteoarthritis limiting ambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Complete a 12-week Exercise Therapy Program | 12 weeks.
  Completion of a 12-week program in the treatment group will be completion of the remote SVS SET Program while the "usual care" group may have an in-person 12-week exercise therapy program.

SECONDARY OUTCOMES:
Mobile Phone Delivered 6-Minute Walk Test | Weeks 0, 6 and 12
  Mobile-phone delivered 6-minute walk test result in steps to be reported at three time points.
Passive Activity as Measured on Mobile Device | 12 weeks.
  Daily passive step count activity as measured by sensors in mobile phone.
Quality of Life Survey as measured by the mini-Walking Impairment Questionnaire (mini-WIQ) | Weeks 1, 6, and 12
  QoL questionnaires will be asked on the mobile phone at three time points.
Adherence as Measured by Completion of Scheduled Daily Walks | 12 weeks.
  Adherence to the recommended exercise therapy frequency (3 walks per week) and duration (for at least 30 minutes or more) will be measured
Freedom From Intervention as Measured by Absence of Surgical Intervention at One Year | 1 year.
  Freedom from any surgical intervention will be reported at one year by performing a chart review.

IPD SHARING:
Plan to Share IPD: No